CLINICAL TRIAL: NCT06463912
Title: Screening for Hepatitis c in People Who Inject Drugs in Armenia-Colombia
Acronym: HCV-PIWD
Status: Recruiting | Type: Observational
Sponsor: Asociación Colombiana de Hepatología (Other)
Responsible Party: Principal Investigator, Diana Rocio Chavez Bejarano, Bacteriologist Clinical Epidemiologist, Asociación Colombiana de Hepatología
Other Study IDs: CO-US-987-7106
Record Dates: First submitted 2024-06-06; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Hepatitis C Virus Infection
Keywords: Hepatitis C chronic; Drug Use; Hepatitis C Antibodies rapid test
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People who inject drugs in Armenia-Colombia: Persons over 18 years who injected drugs (PWID), living in the city of Armenia-Colombia.
  Interventions: Other: Does not apply

INTERVENTIONS:
Other: Does not apply — A descriptive cross-sectional study will be carried out in the city of Armenia-Colombia. A total of 205 PWID, 18 years to 65 years old will be included. They will be selected through the implementation of the respondent-driven sampling (RDS).
  Other Names: Opportunity screening

SUMMARY:
Hepatitis C virus infection is a major cause of chronic hepatitis, cirrhosis, and liver cancer. The risk of developing cirrhosis for people with chronic infection with the virus ranges from 15% to 30% over 20 years. Despite undeniable advances in the treatment of hepatitis C infection and the WHO strategy to eliminate hepatitis C by 2030, this infection continues to be a major public health problem globally and many HCV-positive individuals are unaware of their HIV status. People who inject drugs (PWID) are at increased risk for HCV. Several studies have reported high HCV prevalence rates, especially among PWID. PWID are usually exposed to a higher risk of various infectious diseases, mainly due to their drug consumption behaviors and habits, in addition to the risks and harms associated with the respective routes of self-administration.

Worldwide, there are around 11 million PWIDs and there are approximately 2.3 million coinfections between HIV and HCV worldwide, of which more than half (1.3 million) occur in PWID. The coexistence of these two health conditions leads to accelerate the progression of liver disease. The global prevalence of HCV in 2019 among PWID was 50.2%, which is equivalent to 5.6 million people who inject drugs and live with hepatitis C. PWID had been considered a difficult group to reach, manage, and treat because HCV treatment management in these individuals is challenging and they have a higher risk of reinfection and some past HCV treatment guidelines excluded PWIDs from consideration, citing concerns about adherence, increased susceptibility to side effects, and reinfection. However, there is now compelling evidence that HCV treatment is safe and effective among PWID.

In Colombia, the prevalence of hepatitis C among PWID has been measured locally in some cities. In Bogotá, it went from 1.7% in 2002 to 6.7% in 2014. For 2021, the prevalence of hepatitis C was measured in Bogotá, Medellín, Santiago de Cali, the metropolitan area of Pereira, Dos Quebradas, Medellín, Cucuta, and Armenia. The results of prevalence of antibodies against hepatitis C were as follows: Cali with 80.2%, is the city with the highest reactivity, followed by Pereira and Dos Quebradas with 71.4%, Armenia with 69.6%, and Cucuta with 62.8%. We do not have recent data about the impact of intervention to reduce HVC transmission in those groups.

DETAILED DESCRIPTION:
Research question

¿What is the prevalence of HCV in the PWID in the City of Armenia-Colombia? Through this observational study, the prevalence will be determined by screening PWID for hepatitis C by rapid HCV antibody test, to subsequently perform confirmation with viral load PCR in those seropositive. In addition, support will be provided to patients to facilitate their treatment and linkage to care. The use of a respondent-driven sampling (RDS) method will permit obtaining a statistically valid sample.

The objective of this study is to estimate the prevalence of anti-HCV antibodies in PWID between 18 and 65 years of age in the municipality of Armenia (Quindío) through public health strategies such as screening that allows characterize the affected people and facilitate access to diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 65 years old.
* Having used injected psychoactive substances in the last six months.
* Residing in the city or metropolitan area of study in the last six months.
* Present the invitation coupon.
* Person with Colombian nationality, Venezuelan migrant population.

Exclusion Criteria:

* Person who, due to physical, cognitive, or limitations derived from the use of psychoactive substances, is not able to answer the survey autonomously.
* Be in a state of consumption and is prevented from responding to the survey.
* Refuses to collaborate in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All persons over 18 years who injected drugs (PWID) and live in the city of Armenia- Colombia.
Sampling Method: Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
HCV antibody prevalence rate | 10 months
  Hepatitis C virus prevalence

SECONDARY OUTCOMES:
Proportion of patients with access to HCV treatment | 10 months
  Access to treatment for hepatitis C virus infection

CONTACTS AND LOCATIONS:
Overall Officials: Javier Hernández Blanco, MD, Study Director — Asociación Colombiana de Hepatología
Locations (1):
- Colombian Association of Hepatology, Armenia, Quindío Department, Colombia

IPD SHARING:
Plan to Share IPD: No
Informed consent will be requested in written form to all participants, giving clear and easily understandable information about the objectives of the research. The consent will be explained and doubts about it will be resolved and complete freedom of withdrawal of consent will be given at any time during the study, for the reasons that the subject considers.
  The study will be coordinated by health professionals and the sampling and data collection will be performed by nursing assistants trained in rapid tests. The confidentiality of the data collected will be guaranteed, the information obtained will not be used for purposes other than the current research process, and sensitive data or data that allow the identification of the participating individuals will not be published when the information is disclosed. Not use to use non-public or unpublished Study Data for or in support of any commercial endeavor or use.

DOCUMENTS (1):
  • Study Protocol (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT06463912/Prot_000.pdf